CLINICAL TRIAL: NCT04591795
Title: Efficacy and Safety of Sahastara Remedy Extract Capsules in Treating Primary Osteoarthritis of the Knee Compared With Diclofenac (Clinical Trial Phase II)
Brief Title: Sahastara Remedy Extract Capsule in Primary Osteoarthritis of Clinical Trial Phase II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mr NARIN KAKATUM (Other)
Responsible Party: Sponsor-Investigator, Mr NARIN KAKATUM, Faculty of Medicine, Thammasat University
Organization: Thammasat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-EC-TM-2-116_2/59
Record Dates: First submitted 2019-05-30; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis
Keywords: Sahastara; Osteoarthritis; Herbal Medicine
MeSH Terms: conditions — Osteoarthritis | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 mg SHT extract (Experimental): Drug: Sahastara remedy alcoholic extract comparison with diclofenac
  Interventions: Drug: Diclofenac
- 25 mg dicolfenac (Experimental): Drug: diclofenac comparison with diclofenac
  Interventions: Drug: Sahastara remedy extract

INTERVENTIONS:
Drug: Sahastara remedy extract — The concentration of SHT extract is 100 mg per capsule
  Other Names: SHT extract
  Arms: 25 mg dicolfenac
Drug: Diclofenac — Diclofenac sodium, 25 mg enteric-coated tablets
  Arms: 100 mg SHT extract

SUMMARY:
To study efficacy and safety of Sahastara 95% ethanolic extract capsules compared to treatment Primary osteoarthritis for primary osteoarthritis, it was compared with diclofenac (Phase II).

DETAILED DESCRIPTION:
Sample size 66 volunteers

The patients were divided randomly into 2 treatment groups. The patients in group 1 received the SHT extract 300 mg/day (1 capsule of 100 mg SHT extract three times daily before meals). The patients in group 2 received diclofenac sodium 75 mg/day (1 capsule of 25 mg diclofenac three times daily after meals). In addition, the patients in both groups received 20 mg of omeprazole, 1 capsule before breakfast for protects of Gastrointestinal adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* No pregnancy
* No Serious Medical Condition evaluated by Physical Examination and Laboratory results in 1 month before study
* No Supplementary food and/or Vitamin during the study Able to follow suggestion during the study

Exclusion Criteria:

* Uncontrolled Hypertension (BP>140/90 mm.Hg.) BMI > 30
* Have serious medical condition including Severe peptic ulcer, congestive heart disease, Liver and Renal dysfunction.
* On during use medicine including Rifampicin, Phenytoin, Propranolol, Theophylline

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-13 (Actual); Study Completion 2020-10-13 (Estimated)

PRIMARY OUTCOMES:
Pain score 1 | 28 day
  Pain score from Visual analog scale

SECONDARY OUTCOMES:
Pain score 2 | 28 day
  Pain score from Modified WOMAC score (from Modified Thai WOMAC index)

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Arunporn Itharat, Ph.D., Study Director — faculty of Medicine, Thammasat University
Locations (1):
- Mr. NARIN KAKATUM, Bangkok, BKK, Thailand

IPD SHARING:
Plan to Share IPD: No